CLINICAL TRIAL: NCT03828721
Title: Rx for Success: A Randomized Controlled Trial of Technology-Based Dialogic Reading Training
Brief Title: Rx for Success: RCT of an App for Dialogic Reading Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Reach Out and Read National Office (Unknown); Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-6856
Record Dates: First submitted 2018-03-05; First posted 2019-02-04 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2019-01

CONDITIONS: Literacy; Child Development; Parenting
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled trial involving 2 age categories of low-SES caregiver-child dyads served by the ROR program, each followed for 6 months. For each category, a baseline assessment (pre-) and an outcomes assessment (post-) will be conducted. Category 1 will involve 6 month-old infants, followed until they are 12 months old. Category 2 will involve 18 month-old toddlers, followed until they are 24 months old.
  Families assigned to the control arm in each age category will receive customary ROR, and reading-related developmental surveillance and anticipatory guidance. Control families will also receive a new children's book reinforcing AAP screen-based media recommendations. Families in the intervention arm will receive "enhanced" ROR involving the provision of the Rx for Success (RS) application at the baseline visit (6 months old and 18 months old, respectively).
Who Masked: Participant
Masking Description: Families enrolled in the study will be blinded to its specific aims, other than "We are looking at ways to make reading with children at home more fun and interactive."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - screen time reduction (Active Comparator): Families assigned to the control arm in each age category will receive customary ROR, including the provision of an age-appropriate children's book, and reading-related developmental surveillance and anticipatory guidance. In addition, control families will receive a new children's book reinforcing AAP screen-based media recommendations.
  Interventions: Other: Control - screen time reduction
- Rx for Success Smartphone Application (Experimental): Families in the intervention arm in both age categories will receive "enhanced" ROR involving the provision of the Rx for Success (RS) application at the baseline visit (6 months old and 18 months old, respectively). No additional intervention will take place, other than "push" notifications and other content such as demonstration videos built into the RS application.
  Interventions: Other: Rx for Success Smartphone Application

INTERVENTIONS:
Other: Rx for Success Smartphone Application — The Rx for Success (RS) mobile application (app) was developed by the non-profit, Children, Inc. The app is designed to be informational and motivational with both video and cueing content. The app uses a "View It, Cue It, Do It" model that allows parents to quickly download the smartphone app, view brief videos of age-indexed, research-based language enrichment practices; and regulate a push notification cueing program. Videos embedded in the RS app provide a summary of dialogic reading tailored for the child's age, and suggestions for encouraging verbal interactivity and social-emotional engagement through dialogic reading. Key behaviors reinforced by the app include discussing the story before reading to build interest and enthusiasm, followed by interactive reading modeled by specific types of verbal/behavioral prompts for the parent to make and responses to what the child says or does.
  Arms: Rx for Success Smartphone Application
Other: Control - screen time reduction — Control families will receive a new, specially designed children's book regarding limiting screen-based media use and encouraging healthy/active alternatives (Baby Unplugged: Play, Hutton/Jones, blue manatee press), which lists American Academy of Pediatrics screen time recommendations on the back cover.
  Arms: Control - screen time reduction

SUMMARY:
The purpose of this randomized controlled trial is to explore the efficacy of amplifying dialogic reading training provided to families of infants and toddlers in the ROR program using a novel, smartphone-based application (Rx for Success; RS). The RS app includes videos modeling dialogic reading for a variety of child ages, interactive games, and text messaging reminders to empower parents and other caregivers to increase constructive cognitive and social-emotional stimulation in the home through book sharing. This study addresses an evidence gap regarding the efficacy of dialogic reading training to improve cognitive and social-emotional health using a mobile, technology-based approach. It leverages existing ROR infrastructure and will provide valuable pilot data to improve and scale this inexpensive clinical resource and guide future longitudinal studies, to better serve low-SES, at-risk families.

Aims and hypotheses are as follows:

Specific Aim 1 (Rx for Success; RS): To explore the efficacy of incorporating dialogic reading training via the RS application into ROR during well-child visits for infants (6-12 months old) and toddlers (18-24 months old), compared to standard ROR practice.

Hypothesis 1a (language): Language scores (LENA Snapshot) will be higher in children whose caregivers are provided with the RS app.

Hypothesis 1b (social-emotional): Social-emotional development scores (DECA-I/T items) will be higher in children whose caregivers are provided with the RS app.

Hypothesis 1c (dialogic quality): Dialogic reading quality scores (DialogPR) will be higher in caregivers presented with the RS app.

Hypothesis 1d (attitudes): Attitudes towards shared reading at home (StimQ-I/T items) will be higher in families provided with the RS app.

Specific Aim 2 (exploratory): To explore the effect of providing a smartphone-based app versus a specially designed children's book on screen-based media use.

Hypothesis 2a: Reported screen-based media use (ScreenQ) will be lower in families provided with the RS app, reflecting greater emphasis on interactive shared reading.

Hypothesis 2b: Language (LENA Snapshot) and social-emotional (DECA-I/T items) scores will be higher for children with less reported screen-based media use (ScreenQ).

DETAILED DESCRIPTION:
Shared reading, most often between a parent and child, has been described as "the single most important activity for developing the knowledge required for eventual success in reading." The American Academy of Pediatrics (AAP) recommends daily shared reading beginning as soon as possible after birth. Shared reading occurs in the context of home reading environment, comprised of quantitative factors such as access to books and reading frequency, and qualitative factors such as verbal interactivity and engagement during shared reading. Each of these are addressed by the Reach Out and Read (ROR) program, a population-level, evidence-based intervention based in pediatric primary care clinics. ROR serves low-socioeconomic status (SES) families at-risk for adverse outcomes during a critical span of cognitive, social-emotional and underlying brain development between birth and age 5, when children typically enter kindergarten. The ROR model is for practitioners to capitalize on their privileged access to families with young children during well-child visits to provide a new, age-appropriate children's book, developmental screening related to early literacy skills, and encouragement for families to read together.

Dialogic reading is a method of shared reading that promotes reciprocal dialogue between a caregiver and child, originally developed for low-SES families where such interactivity is often lacking, a major contributor to the widely cited "30-million word gap." The dialogic approach involves specific types of prompts, responses, and references to the child's life, sophistication increasing with age and ability, with the ultimate goal of the child "becoming the reader." Behavioral evidence suggests that dialogic reading may confer moderate to large benefits beginning in infancy, especially in children from low-SES households. These include oral language, narrative comprehension, print concepts, and attention, which are foundational emergent literacy skills. Social-emotional benefits have also been shown, including increased parent-child bonding, pro-social behavior11 and enjoyment of reading. Recent neuroimaging-based studies have also found positive correlation between shared reading quality applying dialogic criteria and brain function supporting emergent literacy in preschool-age children.

A dose-response effect of dialogic reading has been suggested, manifest through greater adherence and practice. However, shared reading quality ("dialogic-ness") tends to be particularly low in low-SES households, attributed to deficient reading abilities, role models, and routines. Several approaches to dialogic reading intervention have been shown to be effective, including video-based training, especially when supplemental instruction and practice are provided to optimize and sustain learning. The ROR program encourages primary care providers to advocate and model dialogic reading during well-child visits, though in practice this can be challenging, given time, reimbursement and other constraints. Thus, despite improved outcomes, there is a need to amplify the ROR intervention in a time-efficient way to address the persistent readiness gap between low-income and more affluent children.

The purpose of this randomized controlled trial is to explore the efficacy of amplifying dialogic reading training provided to families of infants and toddlers in the ROR program using a novel, smartphone-based application (Rx for Success; RS). The RS app includes videos modeling dialogic reading for a variety of child ages, interactive games, and text messaging reminders to empower parents and other caregivers to increase constructive cognitive and social-emotional stimulation in the home through book sharing. This study addresses a major evidence gap regarding the efficacy of dialogic reading training to improve cognitive and social-emotional health using a mobile, technology-based approach. It leverages existing ROR infrastructure and will provide valuable pilot data to improve and scale this inexpensive clinical resource and guide future longitudinal studies, to better serve low-SES, at-risk families.

This is a prospective, randomized controlled trial involving 2 age categories of low-SES caregiver-child dyads served by the Reach Out and Read (ROR) program, each followed for 6 months. For each category, a baseline assessment (pre-) and an outcomes assessment (post-) will be conducted, to explore effects of "enhanced" ROR using the Rx for Success (RS) smartphone app. Category 1 will involve 6 month-old infants, followed until they are 12 months old. Category 2 will involve 18 month-old toddlers, followed until they are 24 months old. Recruitment, informed consent, behavioral testing and intervention will take place at a high-volume primary care clinic based in a major, urban academic medical center in Connecticut (Community Health Center, Inc. at Connecticut Children's Medical Center; CHC@CCMC). Providers in the clinical sites are trained in child development and the administration of ROR during well-child visits between birth and age 5, including those involved with our study at 6, 12, 18, and 24 months old.

Families assigned to the control arm in each age category will receive customary ROR, including the provision of an age-appropriate children's book, and reading-related developmental surveillance and anticipatory guidance. In addition, control families will receive a new children's book reinforcing AAP screen-based media recommendations. Families in the intervention arm in both age categories will receive "enhanced" ROR involving the provision of the Rx for Success (RS) application at the baseline visit (6 months old and 18 months old, respectively). No additional intervention will take place, other than push notifications and other content built into the RS application.

The investigators will recruit 248 children in our 2 age categories: approximately 6 months old (infants, n=124), and approximately 18 months old (toddlers, n=124) via convenience sampling in the CHC@CCMC clinic waiting room during regularly scheduled well-child visits. This study will be powered based on the primary language outcome measure (LENA Snapshot). For a two-group (intervention/control), pre-post repeated-measure analysis with two age categories (6-12 months, 18-24 months), an ANCOVA model will be applied for both age categories and their interaction, to assess the difference in language scores between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestation of at least 34 weeks,
* Age at initial screening 6 months (5.75 months-7.5 months) or 18 months old (17-21 months).
* No documented history of major neurological insult such as intracranial hemorrhage or V-P shunt.
* Comfortable speaking English during their WCC and reviewing/comprehending study materials without a translator, including informed consent.
* Functional literacy in at least one primary caregiver, defined as the ability to navigate the RS application, read prompts provided by the RS application (targeted 6th grade reading level as estimated via the Readable.io website), and understand/provide informed consent, administered in English.
* Possession of a smartphone or tablet device capable of downloading, installing and utilizing the RS application.

Exclusion Criteria:

* Not meeting inclusion criteria above
* Twins

Ages: 6 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Language | 6 months
  Comparison of scores on the LENA Snapshot parent report measure before and after DR intervention between intervention and control groups.
Social-emotional | 6 months
  Comparison of scores on items exerpted from the DECA-I/T Measure, attachment sub scale between intervention and control groups.
Home reading behaviors | 6 months
  Comparison of scores on items exerpted from the StimQ-I/T and DialogPR-IT measures between intervention and control groups.

SECONDARY OUTCOMES:
Screen-based media use | 6 months
  Comparison of ScreenQ scores (screen-based media use at home) between intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Health Center@ Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share this data.

DOCUMENTS (1):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03828721/Prot_000.pdf